CLINICAL TRIAL: NCT04521387
Title: Evaluation of Clinical Efficacy and Comparison of Autologous Platelet Rich Plasma, Hyaluronic Acid, Corticosteroid and Saline Injections for Treating Lateral and Medial Humeral Epicondylopathy
Brief Title: Evaluation of Clinical Efficacy of Different Injection Therapies for Treating Humeral Epicondylopathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DZ-4000-218/19
Record Dates: First submitted 2020-05-21; First posted 2020-08-20 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2021-08

CONDITIONS: Elbow Tendinopathy
Keywords: Tennis elbow; Lateral humeral epicondylopathy; Lateral epicondylitis; injection therapies; platelet rich plasma; hyaluronic acid injection; steroid injection; lateral elbow tendinopathy; epicondylopathia humeri
MeSH Terms: conditions — Elbow Tendinopathy; Tennis Elbow | interventions — Injections; Adrenal Cortex Hormones; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- N1 Platelet Rich Plasma (PRP) (Experimental): 2ml of autologous platelet rich plasma injection
  Interventions: Procedure: injection therapy; Drug: Platelet Rich Plasma
- N2 Corticosteroid (CS) (Active Comparator): 2ml of 7mg Betamethasone injection
  Interventions: Procedure: injection therapy; Drug: Corticosteroid Injection
- N3 Hyaluronic Acid (HA) (Active Comparator): 2ml of 40mg hyaluronic acid with mannitol injection
  Interventions: Procedure: injection therapy; Drug: Hyaluronic Acid Injection
- N4 Saline (NaCl) (Placebo Comparator): 2ml saline (0,9%NaCl) injection
  Interventions: Procedure: injection therapy; Other: Placebo Injection

INTERVENTIONS:
Procedure: injection therapy — The injection will be carried out with aseptic precautions, under regional anesthesia with 1ml of 1% Lignocaine through one puncture of the skin and frequent changes in the inside needle position.
  Other Names: injection
Drug: Platelet Rich Plasma — Platelet rich plasma injection in the painful area of humeral epicondyle.
  Other Names: PRP
  Arms: N1 Platelet Rich Plasma (PRP)
Drug: Corticosteroid Injection — Corticosteroid injection in the painful area of humeral epicondyle.
  Other Names: CS
  Arms: N2 Corticosteroid (CS)
Drug: Hyaluronic Acid Injection — Hyaluronic acid injection in the painful area of humeral epicondyle.
  Other Names: HA
  Arms: N3 Hyaluronic Acid (HA)
Other: Placebo Injection — Saline injection in the painful area of humeral epicondyle.
  Other Names: NaCl
  Arms: N4 Saline (NaCl)

SUMMARY:
Humeral epicondylopathies are common disorders which can significantly impair upper limb function. In case of failure of rehabilitation protocol there is no evidence based second line therapy. It is common practice to perform one of the injection procedures. The biological mechanisms of these procedures are unclear, and may even be contrary. These include, but are not limited to, injections of corticosteroids, autologous platelet rich plasma (PRP) and hyaluronic acid (HA). Despite the frequent use there is much controversy about their clinical effectiveness and more evidence based data are required.

The aim of the study is to compare three different injection therapies for lateral epicondylopathy. In addition, correlation between selected bioactive compounds in PRP and its clinical effectiveness will be evaluated.

The study is planned as a single-center, prospective, randomized, double-blinded, controlled trial on 120 patients aged 30-60 who suffer for lateral epicondylitis. After meeting the inclusion and exclusion criteria patients will receive an injection of leukocyte-rich autologous PRP (N1), corticosteroid (N2), HA (N3) in the area of the common extensors tendon attachment, respectively. Patients from control group (N4) will get an injection of saline in the same area. All groups will be instructed how to perform everyday stretching and strengthening exercises. Evaluation of clinical effectiveness of the treatment will be based on objective measurements such as range of motion, limb girth, grip strength, X-ray and ultrasound examination and subjective measurements such as pain (VAS), functional (PRTEE, DASH, SEV, MEPS) and quality of life questionnaires (SF-36) before and during follow-up period (1, 4, 12, 24, 52 weeks). PRP samples will undergo laboratory analysis of levels of bioactive compounds including platelets, white blood cells, erythrocytes and selected growth factors and inflammatory cytokines.

After data collection, the clinical effectiveness of three different injection therapies will be evaluated and statistically analyzed. Subjective and objective outcomes, safety, costs-effectiveness of three different injection therapies compared to placebo and between each other will be assessed. In addition, correlation between levels of bioactive compounds in PRP and its efficacy will be checked.

DETAILED DESCRIPTION:
The study will be a single-center, prospective, randomized, double-blinded, controlled trial with placebo. It is planned to enroll 120 patients with lateral epicondylopathy and divide them to four equal groups receiving an autologous platelet rich plasma (PRP) (N1=30), corticosteroid (N2=30) or hyaluronic acid (N3=30) injection in the area of lateral epicondyle, or to control group (N4=30) receiving an injection of saline in the same area.

After meeting the inclusion and exclusion criteria and before therapeutic intervention patients will undergo clinical and radiological examination and laboratory analysis of blood samples - complete blood count, C reactive protein (CRP), selected cytokines. Elbow anterior-posterior and lateral view X-ray and ultrasound examination will be performed to find signs of enthesopathy, asses calcifications and to exclude other pathologies.

To measure the clinical effectiveness of the treatment examination including range of motion, limb girth measurements, grip and muscle strength measured by dedicated device (digital dynamometer) and regional pain severity measured by professional digital algometer will be performed. Patients will be asked to fulfil pain, functional and quality of live questionnaires, including Visual Analog Scale for pain intensity evaluation (VAS), Patient-rated Tennis Elbow Evaluation (PRTEE), Disabilities of the Arm, Shoulder, and Hand (DASH), The Mayo Elbow Performance Score (MEPS), The Oxford Elbow Score, The Subjective Elbow Value (SEV) and The Quality of life questionnaire SF-36.

Patients from the experimental group will receive an injection of autologous platelet-rich plasma (PRP) without activator (2ml) in the area of attachment of the common extensor tendon under supervision of ultrasound (N1=30), corticosteroid - 2ml of 7mg Betamethasone (N2=30) or 2ml of 40mg hyaluronic acid with mannitol (N3=30). Patients from control group will get an injection of saline (2ml 0,9% NaCl) in the same area (N=30). The injection will be carried out with aseptic precautions, under regional anesthesia with Lignocaine 1%. Saline injection as placebo intervention for control group was chosen because of a similar impression for the patient comparing to other injections. Also there are some previously reported positive outcomes of that kind of intervention alone. The procedure will be performed in accordance with the principle of double-blinding. Every patient will get identification number which will be randomly assigned to one from all groups, in equal proportion. Both, patient and investigator will not know what kind of substance was used for the treatment. Only person giving the injection will have access to patients identification numbers list and will know the exact type of treatment.

Part of the PRP sample (1ml) will undergo laboratory analysis of levels of bioactive compounds. Assessment of levels and concentrations of platelets, white blood cells and erythrocytes will be performed. The investigators will evaluate the content of selected cytokines in PRP using flow cytometry for growth hormones: Platelet Derived Growth Factor-AA (PDGF-AA), Platelet Derived Growth Factor-BB (PDGF-BB), Vascular Endothelial Growth Factor (VEGF), Epidermal Growth Factor (EGF), Hepatocyte Growth Factor (HGF), Fibroblast Growth Factor basic (FGF), Transforming Growth Factor Beta1 free active (TGFβ1) and inflammatory cytokines: Interleukin-1β (IL-1β), Interferon-α2 (IFN-α2), Interferon-γ (IFN-γ), Tumor Necrosis Factor -α (TNF-α), Monocyte Chemotactic Protein -1 (MCP-1), Interleukin-6 (IL-6), Interleukin-8 (IL-8), Interleukin-10 (IL-10), Interleukin-12p70 (IL-12p70), Interleukin-17A (IL-17A), Interleukin-18 (IL-18), Interleukin-23 (IL-23), Interleukin-33 (IL-33).

Patients will be reassessed 1, 4, 12, 24 and 52 weeks after intervention. All patients will undergo ultrasound examination before treatment and during follow-up period. Every group will be instructed how to perform everyday stretching and strengthening exercises during the whole period of the study. All information about any complications will be collected and evaluated.

After data unblinding, statistical analysis will be performed. Subjective and objective outcomes, safety, costs-effectiveness of three different injection therapies compared to placebo and between each other will be assessed.

There are no original studies comparing clinical effectiveness between corticosteroid, hyaluronic acid, autologous platelet rich plasma and placebo in patients with elbow tendinopathy. There are only few good quality studies on the clinical effectiveness of lateral epicondylopathy treatment with different injection therapies. Most of them compare only one injection method to active comparator or placebo. Usually follow-up period is less than 3 months. Frequent follow-up visits will help to reliably evaluate rate of recurrence and to evaluate correlation between subjective and objective (e.g. USG) findings.

It is believed that results of this study will show significant positive clinical effect of different injection treatments of patients with lateral humeral epicondylopathy. The investigators would like to find which one from injection treatments among corticosteroids, autologous platelet rich plasma and hyaluronic acid will provide best outcomes, safety profile, short and long-term efficacy, cost-effectiveness and the fastest return to work. The results of the study will increase the knowledge about the treatment of lateral epicondylopathy, helping to create a reliable algorithm for supporting the decision-making process in everyday clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* pain on the lateral side of the elbow joint for at least three months,
* confirmation of lateral epicondylitis in at least one provocative test,
* no previous invasive treatment,
* no improvement after rehabilitation

Exclusion Criteria:

* nervous system diseases related to the upper limb,
* hematological diseases,
* diabetes,
* tumors of upper extremity,
* gout,
* advanced osteoarthritis,
* previously performed operations around the elbow joint,
* suspicion of the infectious process,
* pregnant

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain level assessed by Visual Analog Scale | 0, 1, 4, 12, 24, 52 weeks
  the change of pain level in the region of lateral or medial humeral epicondyle after treatment represented on Visual Analog Scale (VAS) scoring from 0 (no-pain) to 10 (worst imaginable pain)
Change in functional outcome assessed by Patient-rated Tennis Elbow Evaluation | 0, 4, 12, 24, 52 weeks
  the change in the results of functional questionnaire - Patient-rated Tennis Elbow Evaluation (PRTEE), scale from 0 to 100, lower value means less disability

SECONDARY OUTCOMES:
Change in muscle strength assessed by hand held dynamometer | 0, 4, 12, 24, 52 weeks
  the forearm muscle strength and grip strength change after treatment measured by hand held dynamometer (higher load means better outcome)
Change in ultrasound examination image | 0, 4, 12, 24, 52 weeks
  any changes in ultrasound examination images of lateral or medial humeral epicondyle region after treatment
Change in results of quality of life questionnaire SF-36 | 0, 4, 12, 24, 52 weeks
  any changes in the results of The Quality of life questionnaire SF-36, scale 0-100, lower score means more disability
Change in functional outcome assessed by Disabilities of the Arm, Shoulder, and Hand | 0, 4, 12, 24, 52 weeks
  the change in the results of functional questionnaire - Disabilities of the Arm, Shoulder, and Hand (DASH), scale from 0 to 100, higher scores reflects to more disability
Change in functional outcome assessed by The Subjective Elbow Value | 0, 4, 12, 24, 52 weeks
  the change in the results of functional questionnaire - The Subjective Elbow Value (SEV), scale from 0 to 100%, subjective self rating of patients elbow, 100% means normal elbow
Change in functional outcome assessed by Mayo Elbow Performance Score | 0, 4, 12, 24, 52 weeks
  the change in the results of functional questionnaire - Mayo Elbow Performance Score (MEPS), scale from 0 to 100, higher value indicates a better condition
Change in functional outcome assessed by The Oxford Elbow Score | 0, 4, 12, 24, 52 weeks
  the change in the results of functional questionnaire - The Oxford Elbow Score, scale from 0 to 100, higher value indicates a better condition

OTHER OUTCOMES:
Rate of adverse events | 0, 1, 4, 12, 24, 52 weeks
  collecting information about any adverse events related with treatment
Comparison of treatment cost-effectiveness | 52 weeks
  comparison of different methods total treatment costs from intervention to complete recovery

CONTACTS AND LOCATIONS:
Overall Officials: Pawel Reichert, PhD, Principal Investigator — Division of Sports Medicine/ Wroclaw Medical University
Locations (1):
- Sport Division, Wroclaw Medical University, Wroclaw, Woj. Dolnośląskie, Poland

IPD SHARING:
Plan to Share IPD: No